CLINICAL TRIAL: NCT00287794
Title: Study on the Quality of Sleep in Patients With Rheumatoid Arthritis
Brief Title: Quality of Sleep in Patients With Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kobe University (Industry)
Responsible Party: Shunichi Shiozawa MD, Kobe University Graduate Scool of Medicine
Other Study IDs: sshiozawah180206
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; sleep disturbance
MeSH Terms: conditions — Arthritis, Rheumatoid; Parasomnias | interventions — Diazepam; Melatonin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples for Western blot for inflammatory cytokines and transcription factors responsible for arthritis.

INTERVENTIONS:
Drug: diazepam, melatonin — Administration of diazepam or such drugs may improve the sleep disturbance of patients with RA.

SUMMARY:
As one of the characteristic clinical features of the patients with rheumatoid arthritis, the unique character of the patients, somewhat difficult to be persuaded but theoretical, has long been pointed out. The investigators hypothesized that this unique character might be due to the sleep disturbance in the patients possibly due to severe pain of arthritis or unique biochemical disease activities. The investigators test (1) the sleep quality of the patients and draw some characteristic features, and (2) investigated the connection between unique biochemical changes such as the increase of c-fos or wee-1.

DETAILED DESCRIPTION:
Under the hypothesis the unique character of patients might be due to the sleep disturbance in the patients possibly due to severe pain of arthritis or unique biochemical disease activities. We do following studies; The study of sleep quality of the patients; The number of patients expected to be included in the study is 1,000. Inclusion criteria is the ACR criteria, and exclusion criteria is any defined disease conditions of sleep disorders in ICSD. The method includes questionnaire using the Pittsburgh Sleep Quality Index (PSQI) scoring and Epworth scoring, and actigraphy measurement for more than 3 days. In a portion of the patients, we measure clinical arthritis activities in conjunction with western blot for c-fos and wee-1 as well as routine clinical laboratory tests. Also in a portion of the patients, we do the polysomnography study; expected number of participants would be 100. We also plan to test the effect of good sloop on arthritis in a portion of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling the American College of Rheumatology criteria of rheumatoid arthritis

Exclusion Criteria:

* Any defined sleep disorders of International Classification of Sleep Disorders (ICSD)

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients with rheumatoid arthritis with or without sleep disturbance.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2006-02; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shunichi Shiozawa, MD, PhD, Study Director — Faculty of Heath Science, Kobe University School of Medicine
Locations (1):
- Konan Kakogawa Hospital, Kakogawa, Hyōgo, Japan

REFERENCES:
- See also: Kobe University Home Page — http://www.kobe-u.ac.jp/